CLINICAL TRIAL: NCT03875521
Title: Impact of the Working Shift Organization on the Caregivers' Satisfaction and Quality of Life at Work, and the Performance of the Intensive Care Units.
Brief Title: Working Shift Organization, Caregivers' Satisfaction and Quality of Life at Work, and Performance.
Acronym: IOTA-REA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17057HLJ
Record Dates: First submitted 2018-12-07; First posted 2019-03-14 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Work-Related Condition
Keywords: Work Schedule Tolerance; Observational Study; Intensive Care Units/manpower; Job Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 12 hours
- < 12hours

SUMMARY:
This is a prospective, non-randomized, multicenter, observational national study, involving centers with different working shift organizations.

Participating centers are 24 French adult intensive care units with different working shift organizations (12-hours shift vs. less than 12-hours shift) in public hospitals.

Caregivers (doctors, nurses and assistant nurses) constitute the population of the study.

The duration of the study is 13 months.

The aim of this study is to evaluate the impact of the working shift organizations on:

* The intensive care units operation;
* The use of outside staff;
* The caregivers' quality of life at work;
* The caregivers' satisfaction at work;
* The nursing work environment;
* Psychosocial and organisational work constraints
* The performance of the intensive care units;
* The costs and efficiency of the working shift organizations.

DETAILED DESCRIPTION:
The critical review of the scientific literature leads us to conclude that there are heterogeneous, and sometimes discordant, results about the impact of a 12-hours working shift organizations on caregivers, hospitals and unit operation, compared with less than 12-hours working shift organizations. This variety and ambiguity of the results could stem from lack of documentation and/or lack of quality of the studies' methodology, the choice of the outcomes, a too short time period for analysis after an organizational change.

In addition, the sociologist analysis is rarely developed. Finally, quite a few studies are declarative, therefore, whatsoever objective outcome is measured.

The determinants of the choice of working shift organization in health facilities are interlinked with multiple factors. Individual and economic factors are considered, as well as clinical risk management, continuity of care and continuity of public services. To the best of our knowledge, no study have evaluated the capacity to maintain a continuity of public health services using 12-hours working shift organization, in particular in French intensive care units subjected to a regulation on nursing and assistant nursing workforce per patient. Besides, there is no data about the impact of 12-hours working shift organization on the performance of intensive care units regarding clinical risk management.

Our hypothesis is that a 12-hours working shift organization may result in a more important number of hours during which the French standard ratio of 1 nurse for 2.5 patients is observed or during which the intensive care beds are not closed, compared with a less than 12-hours working shift organization, with similar caregivers quality of life and performance of intensive care units.

First month of the study: self-administered questionnaires used in order to evaluate nursing work environment (Practice Environment Scale of the Nursing Work Index PES-NWI), caregivers quality of life at work (Nottingham Health Profile NHP, Perceived Stress Scale PSS10 and Hospital Anxiety and Depression Scale HADS) caregivers satisfaction at work (Minnesota Satisfaction Questionnaire MSQ) and psychosocial and organisational work constraints (NWI-EO) will be completed by caregivers (doctors, nurses and assistant nurses).

During the study a sociologist will carry semi-structured interviews on a subset of caregivers from different participating centers.

Eleventh month: self-administered questionnaires used during the first month of the study will be completed again by all caregivers under the same conditions.

One year study period: human resources, activity and performance data will be collected from the beginning to the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* assistant nurses, nurses, doctors
* working in an hospital intensive care unit

Exclusion Criteria:

- opposition to use data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: volunteer caregivers: health care staff of 24 intensive care units will be included in the study: doctors, nurses and assistant nurses
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
intensive care units operation | during 1 year
  Percentage of hours during which the French standard ratio of 1 nurse for 2.5 patients in intensive care units is not observed or during which intensive care beds are closed

SECONDARY OUTCOMES:
use of outside staff | during 1 year
  number of hours during which outside staff is used in participating units (temporary staff, staff working overtime or dedicated supply team staff) during unannounced work stoppages
caregivers' quality of life at work | first and eleventh months of the study
  doctors, nurses and assistant nurses quality of life at work evaluated by using Nottingham Health Profile (NHP)
caregivers' quality of life at work | first and eleventh months of the study
  doctors, nurses and assistant nurses quality of life at work evaluated by using Hospital Anxiety and Depression Scale (HADS)
caregivers' quality of life at work | first and eleventh months of the study
  doctors, nurses and assistant nurses quality of life at work evaluated by using Perceived Stress Scale (PSS10)
caregivers' satisfaction at work | first and eleventh months of the study
  Caregivers' satisfaction at work evaluated with the Minnesota Satisfaction Questionnaire (20-MSQ) and individual interviews with a sociologist.
Nursing Work Environment | During one year
  Evaluated with aggregated data of services (absenteeism rate, delay of recruitment, nurses/patient ratio, assistant nurses/patient ratio, nurses/doctor ratio, assistant nurses/doctor ratio, doctors/patient ratio, number of nurse manager, number of hours worked beyond the expected range, bed occupancy rate, number of days during which beds are unexpectedly closed) and compared between the group of twelve hours working and the less than twelve hours working.
Measure of the performance of intensive care units | during 1 year
  adverse events defined as death in intensive care units (matched to IGS2), and/or adverse events (self-extubation) and/or healthcare-associated infections (bacteremia and sepsis on non-bacteremia catheters)
Budgetary impact | during one year
  The main outcome measure is the total costs (in €) measured by the total labor costs. Labor will be estimated in full-time equivalents, recorded on the time sheets for both medical and non-medical staff.
  The outcome measure is in € and FTEs
psychosocial and organisational work constraints | first and eleventh months of the study
  nurses' and assistant nurses' psychosocial and organisational work constraints evaluated with the Nursing Work Index - Extended Organisation (NWI-EO) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves BLANCHARD, RN, MSN, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- medical-surgical intensive care unit - TENON hospital (AP-HP), Paris, France

IPD SHARING:
Plan to Share IPD: No